CLINICAL TRIAL: NCT00689637
Title: A Single-Centre, Double Blind, Randomized, Two-Way Cross-Over Study of Repeated Doses of AZD3480 and Single Dose of Warfarin to Evaluate the Pharmacokinetic Interaction of AZD3480 and Warfarin and the Effect of AZD3480 Pharmacodynamic in Healthy Male Subjects (Phase I
Brief Title: Drug Interaction Study Between AZD3480 and Warfarin
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans-Göran Hårdemark, MD, PhD, Medical Science Director, AstraZeneca R&D Södertälje, Sweden
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D3690C00014; EudraCt nr 2007-004756-37
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Alzheimer's Disease
Keywords: AZD3480; Warfarin; Drug interaction
MeSH Terms: conditions — Alzheimer Disease | interventions — ispronicline; Warfarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD3480 + warfarin
  Interventions: Drug: AZD3480; Drug: Warfarin
- 2 (Experimental): Placebo+ warfarin
  Interventions: Drug: Placebo; Drug: Warfarin

INTERVENTIONS:
Drug: AZD3480 — AZD3480 capsules qd, 12 days
  Arms: 1
Drug: Placebo — Placebo capsules qd, 12 days
  Arms: 2
Drug: Warfarin — Warfarin: single dose on day 6

SUMMARY:
The purpose of the study is to evaluate if AZD3480 and warfarin interact with each other or not, i.e. show the same or altered plasma concentration profiles when co-administered compared to administered alone.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent
* Clinically normal physical findings and laboratory values

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma within three weeks before the first dose
* History of clinically significant disease
* Use of prescribed medication during the 2 weeks before administration of the first dose of investigational product

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2007-09; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during days 5 and 6

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Göran Hårdemark, MD, Study Director — Clinical Neuroscience TA AstraZeneca R&D Södertälje, Sweden; Cyril Clarke, MD, Principal Investigator — ICON Development Solutions Manchester, UK
Locations (1):
- Research SIte, Uppsala, Sweden